CLINICAL TRIAL: NCT03489993
Title: Interplay of FGF23 and Angiotensin-(1-7) in Hypophosphatemia (GAP)
Brief Title: FGF23 and Angiotensin-(1-7) in Hypophosphatemia (GAP)
Acronym: GAP
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00049606
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-03

CONDITIONS: Hypophosphatemia; X-linked Hypophosphatemia; Renin-angiotensin System; Left Ventricular Hypertrophy
Keywords: FGF23; Angiotensin-(1-7); Hypophosphatemia
MeSH Terms: conditions — Hypophosphatemia; Familial Hypophosphatemic Rickets; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FGF23-Related Hypophosphatemic Diseases: The diagnostic tests Ang II, Ang-(1-7), FGF23, and klotho will be measured in the cohort. Patients in the cohort will have the diseases X-linked hypophosphatemia (XLH), autosomal dominant hypophosphatemic rickets (ADHR), autosomal recessive hypophosphatemic rickets type 1 (ARHR1), autosomal recessive hypophosphatemic rickets type 2 (ARHR2), osteoglophonic dysplasia, Jansen-type metaphyseal chondrodysplasia, Raine syndrome, McCune-Alright syndrome, and epidermal nevus syndrome (ENS).
  Interventions: Diagnostic Test: Ang II and Ang-(1-7); Diagnostic Test: FGF23 and klotho

INTERVENTIONS:
Diagnostic Test: Ang II and Ang-(1-7) — Measured in plasma and urine using radioimmunoassays.
Diagnostic Test: FGF23 and klotho — Measured using ELISA's.

SUMMARY:
Hereditary hypophosphatemia encompasses rare genetic conditions characterized by renal phosphate wasting. Increased circulating levels of fibroblast growth factor 23 (FGF23), a key regulator of phosphorus metabolism, are critical to the pathophysiology of these diseases, most notably in X-linked hypophosphatemia (XLH). Increased FGF23 induces hypertrophy and scarring in the heart in part via stimulating the traditional renin-angiotensin system (RAS) pathway, angiotensin-converting enzyme (ACE)/angiotensin (Ang ll), particularly in patients with chronic kidney disease, but the effect of FGF23 on the heart in patients with FGF23-related hypophosphatemic diseases is unknown. In addition, the relationship between FGF23 and the angiotensin-converting enzyme 2 (ACE2)/angiotensin-(1-7) (Ang-(1-7) pathway of the RAS is unknown.

The objective of this study is to describe the relationship between FGF23, which causes low phosphorus levels, and components of the RAS in the blood and urine to help the investigators understand why the disease occurs and how to better treat it.

Subjects will be identified by querying the Electronic Medical Record according to medical diagnosis. Thirty subjects, 2-24 years of age, will be recruited from the tertiary care Pediatric Endocrinology and Pediatric Nephrology clinics at Brenner Children's Hospital. Inclusion criteria include a confirmed diagnosis of hereditary FGF23-related hypophosphatemia. Clinical data will be obtained from the Electronic Medical Record. Each subject will undergo study assessments at baseline, 6 months and 1 year that include blood work, an echocardiogram, and blood pressure measurements.

The primary hypothesis is that subjects with higher Ang-(1-7) levels have lower rates of cardiac hypertrophy and thus are protected against high FGF23 levels. The secondary hypothesis is that subjects with higher Ang-(1-7) levels have lower systolic blood pressure.

DETAILED DESCRIPTION:
Clinical data will be collected from the Electronic Medical Record, including age, sex, parent-reported race, past medical and family histories, and current medications. The investigators will calculate body mass index and define overweight/obesity as a body mass index ≥85% percentile for age and sex. The investigators will calculate the estimated glomerular filtration rate to measure renal function based on serum creatinine standardized to age, sex, and height.

Blood (less than 5 mL) and urine samples will be collected at each study visit at the same time as routine clinical labs. Ang ll and Ang-(1-7) will be measured in the plasma and urine using radioimmunoassays in a CLIA-certified laboratory within the Hypertension and Vascular Research Biomarker Analytical Core at Wake Forest School of Medicine. The investigators will calculate the ratio of the two peptides and, in the urine, standardize their values to urine creatinine. In the blood, creatinine, calcium, phosphorus, and vitamin D will be collected and in the urine, albumin, calcium, phosphorus, and creatinine will be collected all per standard of care. FGF23 and klotho will be analyzed in the Core via commercially available ELISA's.

All patients receive baseline and, if abnormal, follow-up echocardiograms to evaluate for left ventricular hypertrophy.

Blood pressure will be measured at clinic visits. Because age, sex, and height define normative pediatric values, the investigators will standardize blood pressure with z scores.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hereditary FGF23-related hypophosphatemia

Exclusion Criteria:

* Acquired FGF23-related hypophosphatemia
* Age less than 2 years
* Age more than 24 years
* Inability to provide urine sample

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with hereditary FGF23-related hypophosphatemia will be recruited from the tertiary care Pediatric Endocrinology and Pediatric Nephrology clinics at Brenner Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Left ventricular hypertrophy | 1 year
  Higher Ang-(1-7) levels will be associated with a decreased rate of left ventricular hypertrophy

SECONDARY OUTCOMES:
High blood pressure | 1 year
  Higher Ang-(1-7) levels will be associated with lower systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M South, MD MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalton GD, Xie J, An SW, Huang CL. New Insights into the Mechanism of Action of Soluble Klotho. Front Endocrinol (Lausanne). 2017 Nov 17;8:323. doi: 10.3389/fendo.2017.00323. eCollection 2017. PMID 29250031
- [Background] Faul C, Amaral AP, Oskouei B, Hu MC, Sloan A, Isakova T, Gutierrez OM, Aguillon-Prada R, Lincoln J, Hare JM, Mundel P, Morales A, Scialla J, Fischer M, Soliman EZ, Chen J, Go AS, Rosas SE, Nessel L, Townsend RR, Feldman HI, St John Sutton M, Ojo A, Gadegbeku C, Di Marco GS, Reuter S, Kentrup D, Tiemann K, Brand M, Hill JA, Moe OW, Kuro-O M, Kusek JW, Keane MG, Wolf M. FGF23 induces left ventricular hypertrophy. J Clin Invest. 2011 Nov;121(11):4393-408. doi: 10.1172/JCI46122. Epub 2011 Oct 10. PMID 21985788
- [Background] Gutierrez OM, Wolf M, Taylor EN. Fibroblast growth factor 23, cardiovascular disease risk factors, and phosphorus intake in the health professionals follow-up study. Clin J Am Soc Nephrol. 2011 Dec;6(12):2871-8. doi: 10.2215/CJN.02740311. Epub 2011 Oct 27. PMID 22034506
- [Background] Isakova T, Xie H, Yang W, Xie D, Anderson AH, Scialla J, Wahl P, Gutierrez OM, Steigerwalt S, He J, Schwartz S, Lo J, Ojo A, Sondheimer J, Hsu CY, Lash J, Leonard M, Kusek JW, Feldman HI, Wolf M; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Fibroblast growth factor 23 and risks of mortality and end-stage renal disease in patients with chronic kidney disease. JAMA. 2011 Jun 15;305(23):2432-9. doi: 10.1001/jama.2011.826. PMID 21673295
- [Background] Kinoshita Y, Fukumoto S. X-Linked Hypophosphatemia and FGF23-Related Hypophosphatemic Diseases: Prospect for New Treatment. Endocr Rev. 2018 Jun 1;39(3):274-291. doi: 10.1210/er.2017-00220. PMID 29381780
- [Background] Mitsnefes MM, Betoko A, Schneider MF, Salusky IB, Wolf MS, Juppner H, Warady BA, Furth SL, Portale AA. FGF23 and Left Ventricular Hypertrophy in Children with CKD. Clin J Am Soc Nephrol. 2018 Jan 6;13(1):45-52. doi: 10.2215/CJN.02110217. Epub 2017 Oct 12. PMID 29025789
- [Background] Akimoto T, Yoshizawa H, Watanabe Y, Numata A, Yamazaki T, Takeshima E, Iwazu K, Komada T, Otani N, Morishita Y, Ito C, Shiizaki K, Ando Y, Muto S, Kuro-o M, Kusano E. Characteristics of urinary and serum soluble Klotho protein in patients with different degrees of chronic kidney disease. BMC Nephrol. 2012 Nov 23;13:155. doi: 10.1186/1471-2369-13-155. PMID 23176706
- [Background] de Borst MH, Vervloet MG, ter Wee PM, Navis G. Cross talk between the renin-angiotensin-aldosterone system and vitamin D-FGF-23-klotho in chronic kidney disease. J Am Soc Nephrol. 2011 Sep;22(9):1603-9. doi: 10.1681/ASN.2010121251. Epub 2011 Aug 18. PMID 21852584
- [Background] Drew DA, Katz R, Kritchevsky S, Ix J, Shlipak M, Gutierrez OM, Newman A, Hoofnagle A, Fried L, Semba RD, Sarnak M. Association between Soluble Klotho and Change in Kidney Function: The Health Aging and Body Composition Study. J Am Soc Nephrol. 2017 Jun;28(6):1859-1866. doi: 10.1681/ASN.2016080828. Epub 2017 Jan 19. PMID 28104822